CLINICAL TRIAL: NCT02689544
Title: Acute and Chronic Effects of Static and Dynamic Stretching on Flexibility and Neuromuscular and Functional Performance in Healthy Subjects: a Blinded and Randomized Clinical Trial
Brief Title: Effects of Static Stretching and Dynamic in Flexibility and Performance: Blind and Randomized Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Germanna de Medeiros Barbosa (Other)
Responsible Party: Sponsor-Investigator, Germanna de Medeiros Barbosa, Federal University of Rio Grande do Norte, Universidade Federal do Rio Grande do Norte
Organization: Universidade Federal do Rio Grande do Norte (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1.132.671
Record Dates: First submitted 2016-02-11; First posted 2016-02-24 (Estimated); Last update posted 2016-02-24 (Estimated); Status verified 2016-02

CONDITIONS: Neuromuscular Manifestations
Keywords: exercise muscle stretching; range of motion; dynamometer of muscle strength; electromyography
MeSH Terms: conditions — Neuromuscular Manifestations | interventions — Methods; Muscle Stretching Exercises

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- static stretching (Experimental): Group of 15 volunteers (gSS)
  Interventions: Other: intervention with static stretching
- dynamic stretching (Experimental): Group of 15 volunteers (gDS)
  Interventions: Other: intervention with Dynamic Stretching
- control (Other): Group of 15 volunteers (gC)
  Interventions: Other: Control

INTERVENTIONS:
Other: intervention with static stretching — Members of static stretching group performed three sets of 30 second self hamstring stretch (IT) of both lower limbs, with 30 seconds of rest between sets, totaling 3 minute intervention so.
  Arms: static stretching
Other: intervention with Dynamic Stretching — Each subject contracting antagonist muscle (quadriceps) to the target muscle (hamstring), performing dynamic movements of hip flexion with the knee extended, repeated every 1 second. They amounted to 3 of 30 repetitions completing approximately three minutes of dynamic stretching for each lower.
  Arms: dynamic stretching
Other: Control — The control group volunteers no received intervention
  Arms: control

SUMMARY:
The purpose of this study is analyze the effects, acute and chronic, static and dynamic stretching on flexibility and neuromuscular and functional performance in active, healthy individuals.

Study hypothesis:

1. Static stretching program improves flexibility and reduces neuromuscular and functional performance in active, healthy individuals.
2. Static stretching program improves flexibility and neuromuscular and functional performance in active, healthy individuals.

DETAILED DESCRIPTION:
It is a randomized, blinded clinical trial where the first researcher (P1) was responsible for assessments and reassessments; the second searcher (P2) at randomization and inquiry of the subjects in the intervention protocol and the third investigator (P3) for the statistical analyzes.The research was conducted at the Laboratory of therapeutic practices of the Department of Physical Therapy, Federal University of Rio Grande do Norte (UFRN) and started after the approval of the ethics committee.The sample was recruited by convenience by written disclosure, electronics and personal contact in academies and higher education institutions in the city of Natal / RN. The volunteers were randomly distributed through the electronic site http://www.randomization.com (Code: 21318). Two pieces of information were inserted, namely: the sample size and the number of groups. With this data, the site has generated a specific encoding for each group and distributed the subjects randomly into three groups: static stretching (gAE); dynamic stretching (gAD) and control (gC).

Sample size calculation

For the sample size calculation was used G * Power 3.1.0 software and the procedures followed the recommendations of studies prévios45. Based on a pilot study of four volunteers, it has adopted a power of 0.95, considering a significance level of 5%, a correlation coefficient of 0.5, and 0.25 effect size for both, It calculated a "n" sample of 15 individuals for each group ("n" sample = 45). This analysis was performed to reduce the chance of Type II error and to determine the minimum number of individuals required for this investigation. Thus, the sample size was sufficient to provide 95.5% statistical power.

Procedures and evaluation measures

At first all subjects were recorded in the survey through an evaluation form containing information on identification, weight, height, injury history and physical activity .

After the process of randomization and allocation held by P2, the volunteers underwent the first evaluation (AV1) under the instruction of P1. This evaluation was performed at least 48 hours before the 1st stretching session to prevent possible residual effects of isokinetic and functional testing. Other evaluations AV2, AV3 and AV4, were made immediately after the 1st (acute response) and 10th sessions (acute post elongation) and 48 hours after the last (residual chronic response), respectively, for EAG and GAD. Already the subject of gc were subject only to the four evaluation processes, where the last assessment (AV4) coincided with the time related to the stretching protocol of the experimental groups. Despite receiving the same guidelines of the other groups on the importance of stretching activities routines during the study period the volunteers were told they should not perform stretching in the day-to-day.

All had non-dominant leg (MND) tested for flexibility, neuromuscular performance (muscle latency time and isokinetic performance) and functional performance (functional tests) in all four assessments. The MND was used because it is considered less skilled and more trainable, when compared to the MD46. For their identification was asked which member preferred to kick a bola15. However, during the interventions in the experimental groups (GAE, GAD), both members were elongated, evaluating the pain sensation at the end of each session and at the end of the intervention protocols, sensory perception (pleasure / displeasure) in performing elongation. The day of the period in which prevailed the assessments and reassessments was on afternoon shift.

ELIGIBILITY:
Inclusion Criteria:

* (1) male;

  (2) were aged between 18 and 28 years old;

  (3) Body mass index (BMI) of 21 to 25 kg / m2,

  (4) not be participating in lower limb stretching programs;

  (5) be healthy, according to Physical Activity Readiness Questionnaire (PAR-Q) and perform physical activity (recreational, not competitive level) for at least 3 times a week, according to the International Physical Activity Questionnaire (IPAQ)

  (6) no history of injury or disease in the lower limbs in the last six months, without previous surgery in this segment;

  (7) lack of musculoskeletal, cardiorespiratory and neurological disorders that prevent the completion of the evaluation and treatment protocols;

  (8) is not under the effect of medicines that cause muscle relaxation or that inhibit muscle tonic action

  (9) has ROM limitation (degree of muscle shortening) of at least 15 ° of active extension of joelho21, the non-dominant leg (considering 180 the full extent with hip positioned at 90 ° of flexion).

Exclusion Criteria:

* (1) start stretching practice in daily activities during the study period;

  (2) not perform evaluative and intervention procedures;

  (3) absence of at least one of the sessions of stretching protocol;

  (4) appearance of lesions during the period in which the subject is inserted in the survey;

  (5) withdrawal in the study. Thus, it excluded eight volunteers, three per occurrence of injuries during the study period and five per withdrawal, concluding the study with a total of 45 subjects.

Ages: 18 Years to 28 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2015-06; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Range of Motion | Evaluation of range of motion after one month the application of stretching
  Range of Motion measured by Universal Goniometer

CONTACTS AND LOCATIONS:
Overall Officials: Wouber H Vieira, Prof.Dr., Principal Investigator — Universidade Federal do Rio Grande do Norte